CLINICAL TRIAL: NCT00679523
Title: An Open-Label, Rising Multiple-Dose, Multi-Center Study to Evaluate the Safety and Efficacy of Topically Applied AN2690 5.0% and 7.5% Solution for the Treatment of Adult Subjects With Onychomycosis of the Great Toenail
Brief Title: Safety and Efficacy Study of Subjects With Onychomycosis of the Great Toenail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Karl Beutner, MD, PhD, Anacor Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN2690-ONYC-201 Cohort 1 and 2
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Fungal Nail
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): AN2690 Solution, 5.0%
  Interventions: Drug: AN2690 Solution, 5.0%
- Group 2 (Experimental): AN2690 Solution, 7.5%
  Interventions: Drug: AN2690 Solution, 7.5%

INTERVENTIONS:
Drug: AN2690 Solution, 5.0% — Once daily application for 180 days
  Arms: Group 1
Drug: AN2690 Solution, 7.5% — Once daily application for 180 days
  Arms: Group 2

SUMMARY:
The purpose of the study is to determine the safety and efficacy of 5.0% and 7.5% AN2690 Solution in the treatment of distal, subungual onychomycosis of the great target toenail.

DETAILED DESCRIPTION:
The first group of 30 protocol-qualified subjects will be assigned to Treatment Group 1 and given 5% AN2690 Solution. Provided that there is adequate evidence of clinical safety after two weeks of dosing with 5% AN2690 Solution, a second group of 30 protocol-qualified subjects will be assigned to Treatment Group 2 and given 7.5% AN2690 Solution. A third group of 30 subjects will be enrolled and assigned the highest safe concentration of AN2690 evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Witnessed, signed informed consent approved by Ethics Committee
2. Male or female subjects of any race at least 18 years of age but not older than 65 years of age at the time of screening
3. Subjects with a diagnosis of onychomycosis of at least one great toenail and with a positive KOH wet mount from that nail
4. Onychomycosis involving 20-60% of the affected great toenail as determined by visual inspection after the nail has been trimmed
5. The combined thickness of the distal nail plate and the associated hyperkeratotic nail bed <3 mm
6. Affected great toenail to be treated is capable of re-growth as documented by history or recent observation of at least 2 mm of growth
7. Normal or not clinically significant screening safety labs

Exclusion Criteria:

1. Females of childbearing potential not using a highly effective method of birth control (e.g. implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices) during the study
2. Diabetes mellitus requiring treatment other than diet and exercise
3. Subjects with chronic moccasin type of T. pedis
4. Subjects with a history of having failed any previous topical antifungal therapy for their onychomycosis
5. Subjects unwilling to refrain from the use of nail cosmetics such as clear and or colored nail lacquers from the screening visit until the end of the study.
6. Subjects that have not undergone the specified washout period(s) for the following topical preparations or subjects who require the concurrent use of any of the following topical medications:

   * Topical antifungal applied to the feet (does not include antifungals for treatment of T. pedis during the study): 4 weeks
   * Anti-inflammatories, corticosteroids, topical immunomodulators: 2 weeks
7. Subjects that have not undergone the specified washout period(s) for the following systemic medications or subjects who require the concurrent use of any of the following systemic medications:

   * Corticosteroids (including intramuscular injections): 2 weeks
   * Antifungals for treatment of onychomycosis or any systemic antifungal with known activity against dermatophytes: 24 weeks
   * Systemic immunomodulators: 4 weeks
8. Treatment of any type for cancer within the last 6 months
9. History of any significant internal disease
10. Subjects with a medical history of current or past psoriasis of the skin and/or nails
11. Concurrent lichen planus
12. Subjects who are known to be allergic to any of the test product(s) or any components in the test product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure
13. Nail or anatomic abnormalities of the toe, e.g., genetic nail disorders, primentary disorders, onychogryphosis, trauma to the nail(s) to be treated
14. AIDS or AIDS related complex
15. History of street drug or alcohol abuse
16. Any subject not able to meet the study attendance requirements
17. Subjects who have participated in any other trial of an investigational drug or device within 60 days prior to enrollment or participation in a research study concurrent with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
A calculated endpoint of treatment response at Day 180 comprised of the ISGA, clear nail growth and fungal culture results | Day 180

SECONDARY OUTCOMES:
Mycological and clinical response of "complete responders", "partial responders", and "non-responder". | Days 180

CONTACTS AND LOCATIONS:
Locations (9):
- Mexico (9):
  - Unidad de Investigación en Salud (UIS), Chihuahua City
  - Hospital "Dr. Angel Leaño", Guadalajara
  - Instituto Dermatologico Jalisciense, Guadalajara
  - Centro Dermatologico Pascua, Mexico City
  - CIF-BIOTEC Medica Sur., Mexico City
  - IMIC, Mexico City
  - Hospital Universitario Dr. José Eleuterio González, Monterrey
  - MIRC / OCA Hospital, Monterrey
  - ISSEMYM, Toluca